CLINICAL TRIAL: NCT00027976
Title: A Phase II/III Randomized, Double-Blind, Placebo-Controlled Clinical Trial Of Celecoxib In Subjects With Actinic Keratoses
Brief Title: Celecoxib in Preventing Skin Cancer in Patients With Actinic Keratoses
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000069099; UAB-9833; UAB-NQ401A4009; UAB-NQ49902009; NCI-P00-0161; NCI-P01-0197
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2012-11

CONDITIONS: Precancerous Condition
Keywords: actinic keratosis
MeSH Terms: conditions — Precancerous Conditions; Keratosis, Actinic | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 active arm (Experimental): receipt of active drug
  Interventions: Drug: celecoxib
- Group 2 active arm (Experimental): receipt of active drug
  Interventions: Drug: celecoxib
- group 2 placebo arm (Experimental): receipt of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: celecoxib
  Arms: Group 1 active arm; Group 2 active arm
Drug: Placebo
  Arms: group 2 placebo arm

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of celecoxib may be an effective way to prevent actinic keratoses.

PURPOSE: Randomized phase II/III trial to determine the effectiveness of celecoxib in preventing skin cancer in patients who have actinic keratoses.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare celecoxib vs placebo in terms of preventing the development of new actinic keratoses in patients with actinic keratoses.
* Compare these treatment regimens in terms of inducing regression of actinic keratoses in these patients.
* Determine the safety of this drug in these patients.
* Compare the effect of these treatment regimens on potential surrogate end-point biomarkers in areas of actinic keratosis, sun-exposed skin, and non-sun-exposed skin and correlate these biomarkers with clinical outcome in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral celecoxib twice daily for 9 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo as in arm I. Patients are followed at 2 months after completing treatment.

PROJECTED ACCRUAL: A total of 240 patients (120 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Fitzpatrick skin types I, II, or III
* Sun-damaged skin with 10-40 actinic keratoses on the upper extremities (upper arms, forearms, and hands), neck, face, and scalp combined

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 125,000/mm^3
* Hemoglobin at least lower limit of normal
* No significant bleeding disorder

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 1.5 times ULN
* No chronic or acute hepatic disorder

Renal:

* Creatinine no greater than 1.5 times ULN
* BUN no greater than 1.5 times ULN
* No chronic or acute renal disorder

Gastrointestinal:

* No history of or active inflammatory bowel disease
* No active pancreatitis
* Not diagnosed with esophageal, gastric, pyloric channel, or duodenal ulceration within the past 30 days

Other:

* No history of keloid formation
* No known photosensitivity disorder
* No history of hypersensitivity or adverse reaction to sulfonamides, COX-2 inhibitors, salicylates, or other NSAIDs
* No other condition that would preclude study
* No other medical or psychosocial condition that would preclude study
* No other malignancy within the past 5 years except:

  * Carcinoma in situ of the cervix
  * Curatively excised nonmelanoma skin cancer
  * Stage 0 chronic lymphocytic leukemia
  * Any cancer for which the patient is currently without evidence of disease, has not been treated for tumor within the past 6 months, has no current or planned therapy, and has an expected disease-free survival of at least 5 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 30 days since prior systemic immunotherapy
* No concurrent immunotherapy

Chemotherapy:

* At least 3 months since prior topical fluorouracil (5-FU)
* At least 6 months since other prior topical chemotherapy
* No concurrent topical chemotherapy, including 5-FU
* No other concurrent chemotherapy

Endocrine therapy:

* At least 6 months since prior oral or IV corticosteroids for more than 2 consecutive weeks
* At least 6 months since prior inhaled or nasal corticosteroids for more than 4 weeks duration
* At least 14 days since prior topical corticosteroids
* At least 30 days since prior nasal corticosteroids (except mometasone)
* No concurrent oral or IV corticosteroids for more than 2 consecutive weeks during any 6 month period during study
* No concurrent inhaled or nasal steroids (except mometasone) for more than 4 weeks during any 6 month period during study
* No concurrent hormonal or steroidal therapy, including topical corticosteroids
* Concurrent hormone replacement therapy (e.g., estrogen or thyroid hormone replacement) allowed

Radiotherapy:

* At least 6 months since prior local radiotherapy to areas being studied
* At least 30 days since other prior radiotherapy
* No concurrent radiotherapy, including local radiotherapy to areas being studied

Surgery:

* Not specified

Other:

* At least 30 days since prior cryotherapy to target lesions
* At least 60 days since prior laser resurfacing, dermabrasion, or chemical peels
* At least 30 days since prior investigational medication
* At least 14 days since prior topical alphahydroxyacids (e.g., glycolic acid or lactic acid) or retinoids
* At least 30 days since prior systemic psoralens or retinoids
* At least 30 days since prior treatment for esophageal, gastric, pyloric channel, or duodenal ulcers
* At least 30 days since prior aspirin (more than 100 mg/day), other nonsteroidal anti-inflammatory drugs (NSAIDs) or COX-2 inhibitors at a frequency of at least 3 times per week for more than 2 weeks (except cardioprotective doses of aspirin (no more than 100 mg/day)
* No concurrent systemic psoralens or retinoids
* No concurrent prescription or over-the-counter topical medications to areas being studied (e.g., vitamin A derivatives)
* No concurrent cryotherapy to target lesions
* No concurrent laser resurfacing, dermabrasion, or chemical peels
* No other concurrent investigational medications
* No concurrent fluconazole or lithium
* No concurrent chronic NSAIDs or COX-2 inhibitors (at least 3 times per week for more than 2 consecutive weeks per year)
* Concurrent cardioprotective doses of oral aspirin (100 mg per day or less) allowed
* Concurrent moisturizer/emollient or sunscreen allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Compare celecoxib vs placebo in terms of preventing the development of new actinic keratoses in patients with actinic keratoses. | baseline to 2 months after last dose

SECONDARY OUTCOMES:
Compare these treatment regimens in terms of inducing regression of actinic keratoses in these patients. | baseline to 2 months after last dose
Compare the effect of these treatment regimens on potential surrogate end-point biomarkers in areas of actinic keratosis, sun-exposed skin, and non-sun-exposed skin and correlate these biomarkers with clinical outcome in these patients. | baseline to 2 months after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Elmets, MD, Study Chair — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Irvine, California
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Elmets CA, Viner JL, Pentland AP, Cantrell W, Lin HY, Bailey H, Kang S, Linden KG, Heffernan M, Duvic M, Richmond E, Elewski BE, Umar A, Bell W, Gordon GB. Chemoprevention of nonmelanoma skin cancer with celecoxib: a randomized, double-blind, placebo-controlled trial. J Natl Cancer Inst. 2010 Dec 15;102(24):1835-44. doi: 10.1093/jnci/djq442. Epub 2010 Nov 29. PMID 21115882
- [Derived] Bakshi A, Shafi R, Nelson J, Cantrell WC, Subhadarshani S, Andea A, Athar M, Elmets CA. The clinical course of actinic keratosis correlates with underlying molecular mechanisms. Br J Dermatol. 2020 Apr;182(4):995-1002. doi: 10.1111/bjd.18338. Epub 2019 Sep 11. PMID 31299087